CLINICAL TRIAL: NCT00973908
Title: Probiotics for the Prevention of Antibiotics Associated Diarrhoea and Clostridium Difficile Associated Diarrhoea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Health Service, United Kingdom (Other Government)
Collaborators: Wrightington, Wigan and Leigh NHS Foundation Trust (Other); Ferring Pharmaceuticals (Industry); South London and Maudsley NHS Foundation Trust (Other); North Bristol NHS Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Principal Investigator, Christian Selinger, Coordinating investigator, National Health Service, United Kingdom
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WWL - CDiff Prevention; EUDRACT 2008-005244-16
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Diarrhoea
Keywords: Clostridium difficile associated diarrhoea; antibiotic associated diarrhoea
MeSH Terms: conditions — Diarrhea | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VSL#3 (Active Comparator): Patients will receive one VSL #3 sachets twice a day for the duration of the antibiotic course and for one week after.
  Interventions: Drug: VSL#3
- Placebo (Placebo Comparator): Patients will one placebo sachet twice a day for the duration of the antibiotic course and for one week after.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSL#3 — Patients will o receive one VSL #3 sachets twice a day for the duration of the antibiotic course and for one week after.
  Other Names: Bifidobacterium breve; Bifidobacterium longum; Bifidobacterium infantis; Lactobacillus acidophilus; Lactobacillus plantarum; Lactobacillus paracasei; Lactobacillus bulgaricus; Streptococcus thermophilus
  Arms: VSL#3
Drug: Placebo — Patients will one placebo sachet twice a day for the duration of the antibiotic course and for one week after.
  Other Names: Maltose based Placebo
  Arms: Placebo

SUMMARY:
The investigators aim to investigate whether the routine use of the probiotic formulation VSL#3 co-prescribed with antibiotics reduces the incidence of both Antibiotic associated diarrhoea and Clostridium Difficile associated diarrhoea.

DETAILED DESCRIPTION:
The investigators aim to find out whether VSL#3 can prevent Antibiotic associated diarrhoea and Clostridium Difficile associated diarrhoea when VSL#3 is giving during a course of systemic antibiotics. Patients will be randomized in a 1:1 proportion to receive either one sachet of VSL#3 or a similar looking placebo twice a day. This will be given for the length of the antibiotic course and another week thereafter. Follow-up will last until 28 days after the last antibiotic dose. Patient restarted on antibiotics during follow-up will be restarted on the trial medication and the 28 day follow-up will be recommenced.

This trial has 2 co-primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older
* Hospital inpatients
* On systemic antibiotics for an infection
* Antibiotics started within last 48 hours

Exclusion Criteria:

* Diarrhoea at screening
* Unable to take enteral meds
* Patients on intensive care units
* Severe Immunosuppression (neutropenia, AIDS, congenital immunoparesis, chemotherapy)
* Risk of endocarditis (Artificial heart valves, history of rheumatic heart disease or infective endocarditis)
* Regular consumption of probiotics until 1 week prior to admission
* Acute severe pancreatitis Persistent vomiting (two days or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Development of antibiotic associated diarrhoea | 28 days post last antibiotic dose
Development of Clostridium difficile associated diarrhoea | 28 days post last antibiotic dose

SECONDARY OUTCOMES:
Length of Hospital Stay | 28 days post last antibiotic dose
30-day Mortality | 30 days after initiation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Neil Haslam, Principal Investigator — Wirghtington Wigan and Leigh NHS Trust
Locations (5):
- United Kingdom (5):
  - Royal Albert Edward Infirmary, Wigan, Lancashire
  - Queen Elizabeth Hospital, Woolwich, London
  - Frenchay Hospital, Bristol
  - Hull Royal Infirmary, Hull
  - Weston General Hospital, Weston-super-Mare

REFERENCES:
- [Background] Bergogne-Berezin E. Treatment and prevention of antibiotic associated diarrhea. Int J Antimicrob Agents. 2000 Dec;16(4):521-6. doi: 10.1016/s0924-8579(00)00293-4. PMID 11118872
- [Background] D'Souza AL, Rajkumar C, Cooke J, Bulpitt CJ. Probiotics in prevention of antibiotic associated diarrhoea: meta-analysis. BMJ. 2002 Jun 8;324(7350):1361. doi: 10.1136/bmj.324.7350.1361. PMID 12052801
- [Background] Cremonini F, Di Caro S, Nista EC, Bartolozzi F, Capelli G, Gasbarrini G, Gasbarrini A. Meta-analysis: the effect of probiotic administration on antibiotic-associated diarrhoea. Aliment Pharmacol Ther. 2002 Aug;16(8):1461-7. doi: 10.1046/j.1365-2036.2002.01318.x. PMID 12182746
- [Result] Selinger CP, Bell A, Cairns A, Lockett M, Sebastian S, Haslam N. Probiotic VSL#3 prevents antibiotic-associated diarrhoea in a double-blind, randomized, placebo-controlled clinical trial. J Hosp Infect. 2013 Jun;84(2):159-65. doi: 10.1016/j.jhin.2013.02.019. Epub 2013 Apr 22. PMID 23618760